CLINICAL TRIAL: NCT04362436
Title: A Phase II Assessment of the Safety and Efficacy of TheraSphere® Selective Internal Radiation Therapy (SIRT) in the Treatment of Metastatic (Liver) Neuroendocrine Tumours (NETs)
Brief Title: TheraSphere Selective Internal Radiation Therapy (SIRT) as Treatment for Neuroendocrine Tumours With Liver Mets
Acronym: ArTisaN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 231087
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Tumors; Liver Metastases
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TheraSpheres Selective Internal Radiation Therapy (SIRT) (Experimental): Radiation therapy
  Interventions: Radiation: TheraSpheres Selective Internal Radiation Therapy (SIRT)

INTERVENTIONS:
Radiation: TheraSpheres Selective Internal Radiation Therapy (SIRT) — Single-photon emission computed tomography (SPECT) imaging will assess 99mTc-MAA (MAA being macro aggregated albumin) deposition in the tumour bed to estimate the dose of radiation to tumour and healthy tissue, before administration of TheraSpheres to eligible patients

SUMMARY:
This is an open label study for patients with inoperable metastatic neuroendocrine liver deposits to see whether treatment with Selective Internal Radiation Therapy (TheraSpheres) could lead to improved treatment response rates with acceptable toxicity (minimal serious adverse events reported). This research will also look at the progression free survival and quality of life of the patients who decide to join the study.

DETAILED DESCRIPTION:
Neuroendocrine tumours (NETs) are tumours which arise from cells of the neuroendocrine system, which is the mechanism by which the hypothalamus maintains homeostasis. Neuroendocrine cells secrete hormones, a type of signalling molecule, that play a role in many of the body's different processes including growth and development.

Surgical resection remains the only curative approach to NETs. However, due to non-specific representations, over 50% of NETs are unresectable at diagnosis. Patients with metastatic high grade, poorly differentiated tumours have a median overall survival of 5 months, as compared to 33 months for those with metastatic low or intermediate grade, well differentiated disease. The liver is the most common site for metastasis and is directly correlated to a much poorer prognosis if moderately to poorly differentiated disease is seen, with 5-year survival of 50% less than those without liver metastases.

Current treatment for non-resectable NETs include somatostatin analogues, systematic anti-cancer therapy (with etoposide/carboplatin being the most commonly prescribed regime), radionuclide therapy, Meta-iodobenzylguanidine Therapy (MiBGG) and Peptide Related Radiation Therapy (PRRT). The last showing great promise in clinical trials with progression free survival at 20 months of 65.2% in the Netter1 trial. However, this therapy is reliant on tumoural expression and a key density of the somatostatin 2 receptor (SSTR2), a feature that is often lost with increasing grade and aggressiveness of disease. In short, the current proposed treatments for non-resectable NETs are still to be optimised and depend heavily on patient status, SSTR2 expression and in the case of chemotherapy, is based on evidence of treatment regimens for other types of cancer.

Selective Internal Radiation Therapy (SIRT), by hepatic arterial delivery of yttrium-90 (Y-90) labelled microspheres, is a safe and effective locoregional therapy that combines a dual anticancer therapy, combining the effects of hepatic arterial embolization with targeted delivery of high dose radiation. This selectively delivers a tumouricidal dose of beta-radiation to the liver tumour, while maintaining a low radiation dose to surrounding normal tissue. 20% of the blood supply of healthy liver comes from the hepatic artery, while 90% of liver tumours derive >90% of their blood supply from the same artery and so the hepatic artery is therefore a compelling target to deliver largely tumour specific treatment, sparing healthy liver. SIRT microspheres are also small enough to get trapped in the liver microvasculature but too large to pass through capillary beds and should therefore not reach other places of the body to cause unwanted side effects.

TheraSpheres consist of an yttrium-90 containing glass microsphere. Yttrium-90 is a pure beta emitter with a half-life of approximately 64.1 hours. It has the same toxicity profile as many chemotherapy agents with the common side effects reported as fatigue, anorexia, pain, nausea and vomiting. In a past clinical trial on NETs, SIRT has shown a radiological response rate of 63% and a median survival of 70 months.

ELIGIBILITY:
Inclusion Criteria:

All patients must be discussed at a specialist hepatobiliary multi-disciplinary team meeting (MDT) and meet the following criteria:

* Histologically confirmed neuroendocrine tumour, with documented grade.
* >18 years of age
* Patients may be on SSAs concurrently.Patients must have had at least one previous line of therapy
* Unresectable liver only or liver predominant metastases (typically involving >25% but <60% of the liver, and technically inoperable, or unfeasible secondary to medical comorbidity)
* Have measurable disease by RECIST 1.1 criteria
* Life expectancy of >12 weeks
* Eastern Cooperative Oncology Group (ECOG) / World Health Organisation (WHO) Performance Status of 0-1
* Adequate liver function (bilirubin less than 34 umol/L in the absence of a reversible cause)
* Blood work: patients must have

  * Platelet count of > or = to 50x10^9/L
  * Hb of > or = to 8.5g/dL
  * Alanine Aminotransferase (ALT) and Aspartate transaminase (AST) < 5 x Upper limit of normal (ULN)
  * Serum creatinine < 1.5 x ULN
  * Internal Normalised Ration (INR) < 2.0
* Patients with portal vein thrombosis may be considered, as determined at MDT (A compromised main portal vein as demonstrated on triple-phase CT scan unless selective or super-selective SIRT can be performed and the other safety criteria are fulfilled)

Exclusion Criteria:

Patients who meet any of the following exclusion criteria will NOT be considered eligible for this study.

* Clinically apparent ascites or other signs of hepatic failure on physical examination
* Severe uncontrollable coagulopathy
* No safe vascular access to the liver, as determined by triple phase CT
* Potential for excess radiation exposure (>30Gy) to the lungs, as determined by pretreatment 99mTc-MAA lung shunt (>20% shunt)
* Shunting to the GI tract that cannot be corrected by embolization, as demonstrated by hepatic angiogram
* Previous Transarterial chemoembolization (TACE) or SIRT
* Multiple biliary stents, or ongoing cholangitis, or any intervention for, or compromise of, the Ampulla of Vater
* Previous external bean radiotherapy to the liver
* Systemic anti-cancer therapy within the last 4 weeks (excluding 1st line therapy with SSA)
* Treatment with Vascular endothelial growth factor (VEGF) inhibitors within 3 months prior to therapy
* Previous or concurrent cancer, other than Basal Cell Carcinoma, unless treated curatively 5 or more years prior to entry
* Tumour involvement of >60% of the liver
* Oesophageal bleeding during the last 3 months
* Any history of hepatic encephalopathy
* Transjugular intrahepatic portosystemic shunt (TIPS)
* Must not be at risk of hepatic or renal failure
* Contraindications against angiography
* Pregnancy and breast feeding. Women of child-bearing potential must have a negative pregnancy test 14 days before treatment, and at the time of theresphere administration.
* Subjects with another significant medical, psychiatric, or surgical condition, currently uncontrolled by treatment, which may interfere with completion of the study.
* Must not be participating in concurrent clinical trials evaluating treatment intervention(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Throughout study completion, up to 1 year
  Record incidence of adverse events overall and by severity, as well as serious adverse events using the National Cancer Institute - Common Toxicity Criteria (NCI-CTC) for Adverse Events, version 4.03 (CTCAE V4.03)
Define objective response rate (ORR) | Throughout study completion, up to 1 year
  This is the best overall response (CR+PR) determined by RECIST 1.1

SECONDARY OUTCOMES:
Progression free survival | Throughout study completion, up to 1 year
  Determined by RECIST 1.1 and defined as date of treatment to the date of first documentation of disease progression
Overall survival | Throughout study completion, up to 1 year
  Date of randomisation to the date of death from any cause, or censored at date of last contact
Quality of life | Throughout study completion, up to 1 year
  Evaluated using the European Organisation for Research and Treatment of Cancer (EORTC) questionnaires QLQ-C30 (Quality of Life Questionnaire type C30) at baseline, week 8 and 3 monthly thereafter
Quality of life 2 | Throughout study completion, up to 1 year
  - Evaluated using the European Organisation for Research and Treatment of Cancer (EORTC) questionnaires QLQ-I.NET21 (Quality of Life Questionnaire, type I.Neuroendocrine Tumour number 21) at baseline, week 8 and 3 monthly thereafter

OTHER OUTCOMES:
Radiomics | Throughout study completion, up to 1 year
  Patients will have a liver CT scan at baseline, 12 weeks post SIRT, 3 monthly thereafter and at disease progression - results will be compared to patient clinical data
Measurement of ctDNA, as a biomarker, in response to TheraSpheres | Throughout study completion, up to 1 year
  Blood samples will be collected at screening, week 8, week 12 and at disease progression for ctDNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rohini Sharma, MD, Principal Investigator — Senior Lecturer Medical Oncology and Clinical Pharmacology
Locations (1):
- Imperial College NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sharma R, Slater S, Evans J, Martinez M, Ward C, Izadi H, Wernig F, Thomas R. ArTisaN trial protocol: a single Centre, open-label, phase II trial of the safety and efficacy of TheraSphere selective internal radiation therapy (SIRT) in the treatment of inoperable metastatic (liver) neuroendocrine neoplasia (NENs). BMC Cancer. 2022 Jul 20;22(1):800. doi: 10.1186/s12885-022-09859-9. PMID 35858849